CLINICAL TRIAL: NCT03122249
Title: Use of Telehealth Technologies for Symptom Management Support for People With Advanced Cancer Living in Rural Communities
Brief Title: Oncology Associated Symptoms & Individualized Strategies
Acronym: OASIS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Determined this protocol was not appropriate for ClinicalTrials.gov
Sponsor: Stephanie Gilbertson-White (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor-Investigator, Stephanie Gilbertson-White, Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 201605851
Record Dates: First submitted 2017-02-03; First posted 2017-04-20 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Advanced Cancer
Keywords: Palliative care; Symptom management; Self-management; Rural area; eHealth; telehealth

STUDY DESIGN:
Intervention Model Description: All participants will receive the intervention delivered via the internet
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OASIS (Other): Patients that meet the eligibility criteria will be enrolled in the study and will receive the advanced cancer symptom management intervention
  Interventions: Behavioral: Advanced Cancer Symptom Management

INTERVENTIONS:
Behavioral: Advanced Cancer Symptom Management — For a period of eight weeks patients will use the OASIS web-application daily to help them get better control of their cancer symptoms. In addition, to daily symptom and strategy tracking, participants will have eight e-visits with the nurse-coach via the Zoom application through the UIHC eHealth and eNovation Center to evaluate their progress with managing their symptoms, assess for barriers to implementing strategies, and offering coaching on how to improve symptom management. Questionnaires and blood samples will be collected at baseline (week 0) and follow-up (weeks 4, 8, and 12).

SUMMARY:
Nearly 20% of Americans and 41% of Iowans live in rural or non-metropolitan areas.(1) Lack of access to providers, long travel distances, and a disconnected health system contribute to increased distress and lower quality-of-life (QOL) in people with advanced cancer living in rural areas. (2) In the state of Iowa, 94% of rural residents have high-speed internet access. (3) The University of Iowa Health Care (UIHC) eHealth eNovation Center has developed the infrastructure to address the health care access gap in Iowa. The combination of wide availability of high-speed internet and the eHealth network provides an opportunity to develop and test interventions that leverage this infrastructure in order to address this important palliative care gap.

This is a pilot study to evaluate the feasibility of an eHealth self-management intervention for cancer symptom management. The intervention consists of a web-application that provides tailored educational information about cancer symptoms and a monitoring platform to track symptom distress and strategies used to manage them. Participants will also receive e-visits from a research nurse or research assistant via UIHC eHealth and eNovation video platform. The purpose of this study is obtain feasibility data about the intervention for a future RCT and to evaluate the OASIS intervention with patients living in rural Iowa receiving treatment for advanced cancer. The specific aims are:

1. to evaluate the feasibility of the OASIS intervention to self-manage symptoms of rural patients with advanced cancer, including a) recruitment and retention, b) use patterns, c) usability of each component of the intervention (i.e., the e-visit platform and the web-application), d) acceptability of the intervention and study (i.e., satisfaction, barriers and facilitators to use, burden); and
2. to determine preliminary effects of the intervention on self-management behaviors and symptom severity, symptom distress, and symptom interference.

DETAILED DESCRIPTION:
Overview of study procedures - Participation in the study last for 12 weeks. Phase 1: baseline data collection and orientation to the intervention (week 0); Phase 2: 8 weeks of daily tracking on website and weekly eHealth visits from a nurse and two data collection points (week 4 and week 8); Phase 3: Optional continuation of tracking on website and as needed eHealth visits from a nurse and final data collection (week 12)

Description of the intervention: For a period of eight weeks patients will use the OASIS web-application daily to help them get better control of their cancer symptoms. In addition, to daily symptom and strategy tracking, participants will have eight e-visits with the nurse-coach via the Zoom application through the UIHC eHealth and eNovation Center to evaluate their progress with managing their symptoms, assess for barriers to implementing strategies, and offering coaching on how to improve symptom management. Questionnaires and blood samples will be collected at baseline (week 0) and follow-up (weeks 4, 8, and 12).

Part 1: OASIS web-application. The web-application is a secure web-site developed by The University of Iowa ITS that contains a number of features participants can use to improve their ability to monitor and manage their physical and emotional symptoms. The daily check-in allows participants to keep track of their symptoms and strategies on a day-to-day basis. A data visualization tool provides visual summary of their symptom distress and strategy use over time. A symptom library describes the pathophysiology (in lay language) of 16 common cancer symptoms. A strategy library contains written descriptions and videos of how to implement 47 common symptom management strategies. The contact nurse-coach feature lists the next scheduled coaching visit as well as provides a way to request an extra e-visit sooner if needed. And finally, other resources will provide phone numbers and web links to resources such as the American Cancer Society, the National Cancer Institute, and Patients Like Me. The personal data participants enter into the OASIS web-application is considered level 3 data and will be handled according to The University of Iowa policies and procedure (See X.4 Electronic Records). After baseline data collection, the web-application will guide participants through the web-application to set up their tailored symptom management plan.

Step 1: On the initial login participants will complete an orientation to the intervention that consists of a video and values exercise. The video will briefly describe how physical and emotional symptoms develop during cancer and why symptom management is critically important for patients with advanced cancer. They will then complete a brief values exercise asking them to think about what is important in their lives. The purpose of the values exercise is to help participants make the cognitive connection about how cancer symptoms may be interfering with aspects of their lives they value most.

Step 2: Next the patient will complete a brief profile (first name, age, gender, type of cancer, current cancer treatment) and select an image or avatar for their profile. Going forward computer algorithms that are driven by information provided by the participant will tailor the experience. For example, the cancer ribbon in the OASIS logo will then change to the color associated with their cancer.

Step 3: Participants will then be instructed to select at least one symptom they want to control better. The selected symptoms will be automatically added to the Symptom Tracker feature of the application. The order in which the symptoms are presented on this screen will be based on the answers provided in the profile. The most common symptoms for that cancer and treatment will be presented first at the top of the list based on behind the scenes decision algorithm. On this screen they can simply choose symptoms from the list or read about common cancer symptoms in the symptom library.

Step 4: Next, participants will select at least one symptom management strategy to use for each symptom. Participants can simply select strategies from a list or read more about them in the strategy library. Strategies selected will be automatically added to the Strategy Tracker. For each symptom selected, a list of common symptom management strategies known to be effective for that symptom will be suggested.

Step 5: Once the participant has identified at least one symptom to work on and one strategy to use, s/he can begin tracking. After completing steps 1-5, the Main Page will now show their symptom and strategy trackers. At the end of each day, the participant is instructed to rate the symptom distress they experienced in the previous 24 hours for the symptom(s) they are tracking and whether they used the selected strategy or not.

Step 6: While participants are not required to read/watch all the content in the web-application, they are encouraged to explore the symptom library and strategy library to learn more about cancer symptoms and ways they can better manage them. Exploration will be encouraged with factoids and teasers. Each time a participant logs in, a pop-up window with a symptom management fact or tip will appear. This pop-up will link to the appropriate content page if the participant is interested in learning more. For example, "TIP: Did you know that whenever you adjust your opioid pain medicine, you should also adjust your constipation medicines?"

Part 2: Nurse-Coach. Through weekly visit via Zoom (which is an HIPAA compliant web-conferencing platform), the nurse-coach will provide the ongoing encouragement, support, and accountability that has been identified as critical to behavior change in other chronic illness self-management interventions. The focus of the communications will be to evaluate the patient's symptoms and use of management strategies, as well as coach the patient to identify and address barriers to effectively implementing strategies to manage their symptoms. Prior to each e-visit the participant will be encouraged to think about how well each management strategy is working and what barriers they are encountering with implementing the strategy. The nurse-coach will review the symptom distress scores and use of management strategies with the participant. The nurse-coach and participant will then discuss how well the strategies have been working and any barriers s/he has encountered. Reviewing the tracker data and evaluating effectiveness and barriers of the strategies is theorized to help the participant connect the dots between how they are feeling and what they can do to improve their symptom management. The nurse-coach may suggest other strategies to consider, assess if there are underlying symptoms that need to be addressed in order to effectively manage symptoms (such as pain that is causing disturbed sleep), and finally, and/or determine additional medical management is appropriate (such as messaging the physician to change a prescription). The nurse-coach is a key feature of the intervention in that s/he will provide primary palliative care as well as promote a sense of therapeutic working alliance with the patient. For the purpose of fidelity monitoring, the e-visits will be audio recorded using the secure audio recording feature in the Zoom application. Recordings will be transcribed verbatim. Participants will be informed that the e-visits is being recorded. The participants will be notified before the recording begins.

Questionnaires: A member of the research team will assist the patient in completing the questionnaires at the clinic at the time of enrollment. In week 4, 8, and 12 patient will complete questionnaires electronically. They will receive these questionnaires via a Qualtrics survey link through email. The questionnaires take approximately 30-90 minutes to complete. The questionnaires include sociodemographics, usability and acceptability of the intervention, plus instruments evaluating social support, perceived stress, optimism, illness/symptom appraisal, symptom burden, self-management behaviors, coping, and communication with health care provider.

Blood: The patient will be met at the phlebotomy clinic for scheduled blood draws. Blood samples for cytokines will be obtained at the same time as other scheduled blood draws to minimize additional needle sticks. 30 mL of blood will be collected from a central venous access device or using standard venipuncture techniques with sodium heparin and EDTA tubes immersed in an ice bath within 15 minutes. Study personnel will confirm that the patient has not smoked or ingested caffeine for at least one-half hour prior to blood collection. The blood collection takes about 15 minutes.

The entire survey data collection will take 45 to 105 minutes per visit(total for visits is 180 to 420 minutes). Daily use of the web-application for a minimum of 10 minutes is expected, totaling 560 minutes. A total of 12 hours and 30 minutes to 16 hrs and 30 minutes of data collection is expected for the whole study.

Medical record review: Medical records will be reviewed at each study visit via EPIC Care Everywhere for information about cancer type and stage, cancer treatments, co-morbid conditions, clinical blood lab values, and symptom treatment interventions.

The study population consists of 40 adults (18 years or older) that will be recruited at the McCreery Cancer Center Clinic sites in Fairfield, IA and Ottumwa, IA. There is no control group in this study. All participants will receive the intervention. Approximately 1 patients per week are seen at the McCreery Cancer Center that meet eligibility criteria. The investigators plan to approach all eligible participants. With a 50% recruitment rate and expect to reach the sample size within 10 months.

Eligible patients will be identified by the McCreery Cancer Center clinic staff (e.g. nurses, radiation therapists, and oncologists) weekly for the upcoming week. A research assistant will be at the McCreery Cancer Center on day of the scheduled appointment. The clinic staff will ask the patient if they are interested in the study. If the patient agrees, a trained research assistant will confirm eligibility, describe participation, and obtain informed consent. If the patient is interested in participating in the study but unwilling or unable to complete the questionnaires or symptom and strategy tracking on the website, they can have a caregiver assist them. The caregiver will function only as a recorder of the patient's responses and not provide their own perceptions. If the patient is not able to verbally interact with the caregiver to complete the questionnaires or symptom and strategy tracking, then they will not be eligible to participate (or will be dropped from the study if already in the intervention phase).

This intervention is based on patient's ability to perform self-care actions with the use of web-application. Self-management activities is highly dependent on decision making ability. As a reason, if their physical or psychological status deteriorate due to their advanced cancer they will no longer will be able to perform self-management actions nor use the web for self-management and will be excluded from the study. If patient's capacity to consent changes over the course of study, their study participation will end early. The UCSD Brief Assessment of Capacity to Consent will be used to reassess capacity as needed during the study.

This project involves research on DNA. Analyses of associations among genetic markers for cytokine, cancer symptoms, and coping behaviors. DNA samples will be identified and labeled with a unique study ID number. The DNA samples and plasma for cytokine analyses will be labeled with only the study ID and date of collection and kept in a -80º C freezer in a locked in the College of Nursing, Office of Nursing Research. Data from the analyses will be securely stored in RedCap.

Data management and analysis will be the primary responsibility of the PI. Questionnaires and biological specimens will be coded to remove all direct personal identifiers. The code list will be kept in a locked cabinet and secure location, separate from where the questionnaires and specimens are stored. The original consent and screening forms will be stored in a locked cabinet in the project area, separate from any data sources.

These de-identified DNA samples or data may be shared in the future with other researchers studying cancer symptoms and cytokines. Prior to sharing any data, an approved IRB protocol and/or material transfer agreement will be obtained.

SAS 9.3 will be used for all analyses. Initial analysis will involve calculating descriptive statistics for all variables at all study points compared to controls. Outliers will be investigated for accuracy. Patterns of missing data will be examined. Graphical representation of the data will be created and examined at each point and longitudinally. The distributions of variables will be evaluated for normality and homogeneity of variance, and appropriate transformations will be applied as needed or statistical analyses for non-normal data will be utilized. Correlations among variables will be examined. A significance level of .05 will be used for statistical tests.

To evaluate the acceptability and usability of the intervention, multiple components of the study will be examined, including resources and time spent on the intervention for each participant, patterns and sources of missing data. In addition the investigators will review the recruitment procedures, as well as any potential experimental confounders and logistical challenges. Descriptive statistics will be employed for analysis of continuous variables and qualitative analyses will be employed for open-ended questions. This information will be used to refine the OASIS intervention and develop procedures for a pilot RCT in future

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 yrs or older) with a current diagnosis of advanced cancer of solid tumor (stage 3 or 4) origin considered incurable by the treating oncologist,
* Experiencing with at least one distressing symptoms (rated 3 or greater on 0-10 numeric rating scale for symptom distress),
* Able to read and write in English
* Have a laptop, mobile phone and/or tablet with a video camera that can use to access the internet
* Have high-speed internet connection in his/her home

Exclusion Criteria:

* Patients who are not able to complete the study surveys (alone or with assistance) due impaired mental, cognitive, or physical status.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-03-10 (Actual); Primary Completion 2019-01-20 (Actual); Study Completion 2019-09-20 (Actual)

PRIMARY OUTCOMES:
Measuring change in Health Education Impact Questionnaire (heiQ) | Week 0,4, 8, 12
  An outcomes and evaluation measure for patient education and self-management interventions for people. This scale is assessing change between four time points
Measuring change in Symptom burden (MDASI - core) | Week 0,4, 8, 12
  Assess patient-reported symptom severity and interference in patients with cancer. This scale is assessing change between four time points
Measuring change in QOL (FACT-G) | Week 0,4,8,12
  This is a patient-reported outcome measure used to assess health-related quality of life in patients undergoing cancer therapy. This scale is assessing change between four time points.

SECONDARY OUTCOMES:
Recruitment | Week 0
  The number of patients approached who agree to participate
Retention rates | Week 0
  The number of patients who complete measures at each time point
Retention rates | Week 4
  The number of patients who complete measures at each time point
Retention rates | Week 8
  The number of patients who complete measures at each time point
Retention rates | Week 12
  The number of patients who complete measures at each time point

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Gilbertson-White, PhD, Principal Investigator — University of Iowa College of Nursing
Locations (1):
- McCreery Cancer Center, Fairfield, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] U.S. Census Bureau. Urban, Urbanized Area, Urban Cluster, and Rural Population, 2010 and 2000: United States. 2010; https://www.census.gov. Accessed 12/23/2015.
- [Background] Pedro LW, Schmiege SJ. Rural living as context: a study of disparities in long-term cancer survivors. Oncol Nurs Forum. 2014 May;41(3):E211-9. doi: 10.1188/14.ONF.E211-E219. PMID 24769604
- [Background] Connect Iowa. Broadband Infrastructure at a State and Local Level in Iowa. 2015.